CLINICAL TRIAL: NCT03965078
Title: Epiretinal Membrane and Acute Pseudophakic Cystoid Macular Oedema: A Prospective Multi-centre Observational Study of Implications and Treatment outComes
Brief Title: Epiretinal Membrane and Cystoid Macular Oedema Post-cataract Surgery
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: EPIC1
Record Dates: First submitted 2018-07-13; First posted 2019-05-28 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-06

CONDITIONS: Pseudophakic Cystoid Macular Oedema; Epiretinal Membrane
Keywords: cataract surgery
MeSH Terms: conditions — Epiretinal Membrane | interventions — Ophthalmic Solutions; Anti-Inflammatory Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CMO without epiretinal membrane: Subject diagnosed with CMO within 12 weeks of cataract surgery without evidence of epiretinal membrane at the time of diagnosis.
  Interventions: Drug: topical (eye drop) anti-inflammatories
- CMO with epiretinal membrane: Subject diagnosed with CMO within 12 weeks of cataract surgery with evidence of epiretinal membrane at the time of diagnosis.
  Interventions: Drug: topical (eye drop) anti-inflammatories

INTERVENTIONS:
Drug: topical (eye drop) anti-inflammatories — Initial treatment with topical anti-inflammatory eye drops at the discretion of the reviewing clinician

SUMMARY:
This study examines whether the presence of an epiretinal membrane affects the time to resolution, requirement for non-topical treatment, and outcome of pseudophakic cystoid macular oedema.

DETAILED DESCRIPTION:
Cataract surgery is the most frequently performed surgery in the NHS. Cystoid macular oedema (CMO, inflammation and fluid accumulation in the central retina) is the most common visually significant complication following cataract surgery occurring in 1-2% of cases. Many cases resolve with topical anti-inflammatory eye drops. However some cases do not respond and require more invasive treatment modalities eg injections into the eye. If CMO remains persistent this can lead to permanent visual loss. There is little current knowledge on what factors lead to persistence in some cases compared to others. Epiretinal membrane (ERM, a fibrocellular membrane that can form on the inner retina) can be associated with a similar cystoid macular oedema that often does not resolve until the ERM is removed surgically. This study aims to look at whether the presence of an ERM affects how long it takes for cystoid macular oedema to resolve following cataract surgery and the requirement for non-topical treatment modalities.

A prospective, non-interventional, observational study design is proposed. Eligible participants would be identified at one of several participating NHS hospitals in the Wessex Deanery. Subjects with evidence of CMO post-cataract surgery and commenced on treatment would be included. Treatment choice is at the discretion of the reviewing clinician and independent of the study protocol. Investigations performed would be only those conducted as part of standard care. Presence of epiretinal membrane would be determined from review of the medical records. Case- records of eligible participants would be reviewed over a 12-month period to assess response to treatment and type of treatment(s) used. Based on current surgical data recruitment would be estimated to take 18 months to achieve the 165 eligible participants to achieve statistical power.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged 18 years or above.
2. Clinical diagnosis of visually significant pseudophakic CMO in ipsilateral eye within 12 weeks of cataract surgery.

   * The clinical diagnosis needs to be made by an ophthalmologist of Grade ST3 or higher.
   * Visually significant is defined as best recorded visual acuity 6/9 Snellen or worse (or LogMAR equivalent)
3. An OCT has to have been undertaken and needs to show the presence of intra-retinal cysts and OCT thickness (central subfield CSF) outside normal parameters as defined by Grover et al [12] and Wolf-Schnurrbusch at al [13] (For clarity the OCT examination does not need to be undertaken on the same day as the clinical diagnosis of pseudophakic CMO. Any OCT examination undertaken after cataract surgery to the ipsilateral eye within the treatment period showing these characteristics will be acceptable to substantiate the clinical diagnosis of pseudophakic CMO.
4. Started on treatment for cystoid macular oedema
5. Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

The participant may not enter the study if there is evidence that macular oedema may have been present pre-operatively. This will include ANY of the following:

* Evidence of pre-existing macular fluid/oedema
* Active proliferative diabetic retinopathy
* Diabetic macular oedema requiring treatment in the last 2 years
* Active uveitis at the time of cataract surgery
* Neovascular age-related macular degeneration
* Active retinal vein occlusion (branch or central) as evidenced by the presence of retinal haemorrhages at the time of cataract surgery or at time of diagnosis of CMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cystoid macular oedema (CMO) within 12 weeks of undergoing cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Time to resolution of CMO after commencing treatment | 1 year
  The time to resolution of the CMO will be calculated from the time of commencement of treatment until the documented time of resolution (based on clinical entry and confirmation on OCT scan). The clinical notes will be accessed at 3 months, 6 months and 12 month time-points to extract this data from the intervening clinical visits. The patient will complete the study either once the CMO is determined to have resolved or at 12 months post-commencing treatment, whichever is sooner.

SECONDARY OUTCOMES:
proportion of CMO cases that resolve within 3-, 6-, and 12-months | 3, 6 and 12 months
proportion of CMO patients requiring non-topical treatment | 12 months
  To describe the proportion of CMO patients requiring non-topical treatment, to compare this proportion between patients with and without ERM, and to describe the types of treatment received
Visual Acuity | 12 months
  To determine visual outcomes for patients with pseudophakic CMO and to compare these between patients with and without ERM

CONTACTS AND LOCATIONS:
Overall Officials: Yit Fung Yang, Study Director — Portsmouth Hospitals Trust
Locations (1):
- Portsmouth Hospitals Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No